CLINICAL TRIAL: NCT00878033
Title: Autonomic Dysfunction and Inflammation in Chronic Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Matthias Girndt, Prof. Dr. med. habil. Matthias Girndt, Director, Martin-Luther-Universität Halle-Wittenberg, Dept. of Internal Medicine II, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKH-KIMII-001-09
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Autonomic Dysfunction; Chronic Renal Failure
MeSH Terms: conditions — Primary Dysautonomias; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum Samples will be frozen for later Cytokine Sampling.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Diabetic Dialysis Patients
- 2: Non-Diabetic Dialysis Patients
- 3: Healthy Controls

SUMMARY:
This study investigates the relationship between autonomic dysfunction and chronic inflammation in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease Stadium KDIGO 5D for at leat 3 months on Dialysis
* Age >18 years
* Sinus action in EKG
* Patient capable for informed consent
* Written and signed informed consent

Exclusion Criteria:

* Clinical overt signs of infections of any kind
* Active malign disease
* CRP levels above 50 mg/L
* Cardiac Pace Maker
* Atrial Fibrillation
* Refusal of informed consent
* Cardiac Transplantation
* Immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic and Non-diabetic Dialysis Patients. Healthy Controls.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Girndt, M.D., Principal Investigator — University Hospital Halle, Dept. of Internal Medicine II
Locations (1):
- Martin-Luther-Universität Halle-Wittenberg, Dept. of Internal Medicine II, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Derived] Seibert E, Zohles K, Ulrich C, Kluttig A, Nuding S, Kors JA, Swenne CA, Werdan K, Fiedler R, Girndt M. Association between autonomic nervous dysfunction and cellular inflammation in end-stage renal disease. BMC Cardiovasc Disord. 2016 Nov 3;16(1):210. doi: 10.1186/s12872-016-0385-1. PMID 27809785